CLINICAL TRIAL: NCT03040830
Title: Does the Time of Starting Progesterone (P4) Luteal Support (LS) Affects Embryo Transfer (ET) in Long Agonist Protocol Down-regulated ICSI Cycles?
Brief Title: Effect of Timing Progesterone Luteal Support on Embryo Transfer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura Integrated Fertility Center (Other)
Responsible Party: Principal Investigator, Mohamad Elsaid Ghanem, Professor, Mansoura Integrated Fertility Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P4 luteal support and ET
Record Dates: First submitted 2017-01-30; First posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Progesterone Luteal Support in ICSI; Embryo Transfer

STUDY DESIGN:
Intervention Model Description: Double blind Randomized Controlled Trial : the clinicians and the patents were blinded of the allocation group.
  A total of 137 embryo transfers (ETs) were randomly allocated into either group A (67 ) starting luteal support as daily intra muscular (IM) injections of 100 mg prontogest on day of egg retrieval, or group B (66) starting the same P4 dose on day of embryo transfer.Transfer technique was blind tactile using Labotect catheter and was considered difficult if the inner ET catheter was blood stained and /or sounding or dilating the cervix was needed. Cervical traction or blood staining of outer sheath did not indicate difficulty
Who Masked: Participant, Care Provider
Masking Description: The randomization
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Egg retrieval arm (Experimental): 67 ICSI cases are started daily 100 mg IM prontogest on the day of egg retrieval until the day of pregnancy test.
  Interventions: Drug: Progesterone 100 IM/day
- Embryo transfer arm (Active Comparator): 66 ICSI cases are started daily 100 mg IM prontogest on the day of embryo transfer until the day of pregnancy test.
  Interventions: Drug: Progesterone 100 IM/day

INTERVENTIONS:
Drug: Progesterone 100 IM/day — Progesterone IM 100 mg /day was started on day of egg retrieval in egg retrieval arm and on day of embryo transfer in the embryo transfer arm

SUMMARY:
The study aims to know whether starting progesterone luteal support in intra cytoplasmic sperm injection (ICSI) cycles on the day of ovum pickup affects the degree of difficulty of embryo transfer compared with starting luteal support on day of embryo transfer

DETAILED DESCRIPTION:
Double blind Randomized Controlled Trial (RCT) : the clinicians and the patents were blinded of the allocation group.

A total of 137 embryo transfers were randomly allocated into either arm I (67 ) starting luteal support as daily IM injections of 100 mg prontogest on day of egg retrieval , or arm II (66) starting the same P4 dose on day of embryo transfer

ELIGIBILITY:
Inclusion Criteria:

* first ICSI trial, normal uterus, normal cervix, normal ovarian response ,easy mock transfer,patient consenting

Exclusion Criteria:

* age over 38, difficult mock transfer, low and high ovarian response, patient not consenting

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — infertile females undergoing first ICSI cycle
Enrollment: 150 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
difficult embryo transfer | 3 minutes
  presence of blood on embryo transfer catheter and or need for sounding or dilating the cervix to pass the embryo transfer catheter to the endometrial cavity

SECONDARY OUTCOMES:
cycle outcome | 4 weeks
  clinical cycle pregnancy rate calculated as number of clinical pregnancies (gestational sacs shown by ultrasound ) per 100 cases transferred multiplied by 100.Implantation rate calculated by the outcome of dividing the total number of gestational sacs in the arm by the total number of embryos transferred.

REFERENCES:
- [Background] Mochtar MH, Van Wely M, Van der Veen F. Timing luteal phase support in GnRH agonist down-regulated IVF/embryo transfer cycles. Hum Reprod. 2006 Apr;21(4):905-8. doi: 10.1093/humrep/dei437. Epub 2005 Dec 22. PMID 16373409
- [Background] Senciboy D.N and Sharpe-Timms K.L: Progesterone affects the cervix prior to embryo transfer. , Fertility and Sterility ,2001: 76 , Issue 3 , S220 - S221
- [Background] Ghanem ME, Ragab AE, Alboghdady LA, Helal AS, Bedairy MH, Bahlol IA, Abdelaziz A. Difficult embryo transfer (ET) components and cycle outcome. Which is more harmful?. Middle East Fertility Society Journal. 2016 Jun 30;21(2):114-119
- [Derived] Ghanem ME, Bedairy MH, Shaaban A, Albahlol IA. Does the Time of Starting Progesterone Luteal Support Affect Embryo Transfer in Long Agonist Protocol Downregulated ICSI Cycles? A Randomized Controlled Trial. Reprod Sci. 2021 Mar;28(3):897-903. doi: 10.1007/s43032-020-00309-0. Epub 2020 Sep 9. PMID 32909190